CLINICAL TRIAL: NCT00036205
Title: Open-Label, Long Term, Flexible Dose Study Of Safety, Tolerability, And Therapeutic Response In Patients With Parkinson's Disease.
Brief Title: Open Label Sumanirole Study of Safety, Tolerability, and Therapeutic Response In Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M27600011
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — U 95666E

INTERVENTIONS:
Drug: sumanirole

SUMMARY:
The primary objective is to assess the long term safety and tolerability of sumanirole as measured by safety labs, ECG monitoring, vital signs, and adverse event reports in subjects with Parkinson's Disease who participated in previous sumanirole studies.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Modified Hoehn and Yahr Scale Stages 1-4
* Age over 30 years
* Previous participation in prior sumanirole studies

Exclusion Criteria:

* Use of dopamine agonist medications and other medications in defined timeframe
* Unstable dose of CNS active therapies (eg, hypnotics, antidepressants, anxiolytics) within the last 30 days
* Atypical Parkinson's syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases
* Dementia
* History of active epilepsy within the past year
* Significant liver disease with defined laboratory criteria
* Significant renal disease with defined laboratory criteria
* Certain cardiac conditions
* Electroconvulsive therapy in the previous 90 days
* Subjects participating in other drug studies or receiving other investigational drugs within previous 30 days
* Positive pregnancy test at Screen
* Unwillingness to use adequate contraceptive methods
* Lactating women
* History of stereotaxic brain surgery
* Malignant melanoma or history of treated melanoma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984
Dates: Start 2000-08; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary objective is to assess the long term safety and tolerability of sumanirole by measuring Safety labs, ECG monitoring, vital signs and adverse events, over a period of up to 4 years.

SECONDARY OUTCOMES:
Pharmacoeconomics, quality of life, and the long term therapeutic response associated with sumanirole by using Parts II and III of the UPDRS (Unified Parkinson's Disease Rating Scale).
Part II -- Activities of Daily Living, will be collected in order to record the patient's level of function between visits.
Part III will be used to evaluate motor function.
Three quality of life instruments will be employed: a general scale--the Functional Status Questionnaire, a disease specific scale--the Parkinson's Disease Questionnaire, and a utility scale--the EuroQol.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (110):
- United States (103):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Luis Obiapo, California
  - Pfizer Investigational Site, Sunnyvale, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Fairfield, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Trumbull, Connecticut
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lenexa, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Elkridge, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Bingham Farms, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Traverse City, Michigan
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Golden Valley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, Salisbury, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Mount Vernon, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Canfield, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Wenatchee, Washington
  - Pfizer Investigational Site, Marshfield, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (4):
  - Pfizer Investigational Site, Buenos Aires, Barcelona
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Mar del Plata, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogotá, D.C.
- Pfizer Investigational Site, Carolina, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=M27600011&StudyName=Study+of+Safety%2C+Tolerability%2C+and+Therapeutic+Response+In+Patients+With+Parkinson%27s+Disease+With+Sumanirole